CLINICAL TRIAL: NCT03683446
Title: Trends and Outcomes in Laparoscopic Versus Open Surgery for Rectal Cancer From 2005 to 2016 Using the ACS-NSQIP Database, a Retrospective Cohort Study
Brief Title: Trends and Outcomes in Laparoscopic Versus Open Surgery for Rectal Cancer
Acronym: NSQIPc
Status: Completed | Type: Observational
Sponsor: Catherine H. Davis, MD (Other)
Responsible Party: Sponsor-Investigator, Catherine H. Davis, MD, Principal Investigator, Houston Methodist Hospital Physician, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00014677
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Adenocarcinoma; Colorectal Surgery
Keywords: Colorectal Cancer; Colorectal; Colorectal surgery; Surgical complications; Rectal; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic Rectal Surgery: A minimally invasive surgery and specialized technique for performing surgery using smaller incisions (or ports) to enter into the abdomen or anus for a tubular instrument(trochar), and a special camera (laparoscope), which is passed through the trochars to visualize the colon. For abdominal entry, at the beginning of the procedure, the abdomen is inflated with carbon dioxide gas to provide a working and viewing space for the surgeon. For both, the laparoscope transmits images from the abdominal cavity or anus to high-resolution video monitors to allow the surgeon detailed images of the abdomen on the monitor.
  Interventions: Procedure: Laparoscopic rectal surgery
- Open Rectal Surgery: Surgery performed through a single long incision (cut) in the abdomen (belly) to access the colon and/or the rectum.
  Interventions: Procedure: Open rectal surgery

INTERVENTIONS:
Procedure: Laparoscopic rectal surgery — Minimally invasive surgery and specialized technique for performing surgery using smaller incisions (or ports) to enter into the abdomen or anus for a tubular instrument(trochar), and a special camera (laparoscope), which is passed through the trochars to visualize the colon.
  Groups: Laparoscopic Rectal Surgery
Procedure: Open rectal surgery — Surgery performed through a single long incision (cut) in the abdomen (belly) to access the colon and/or the rectum.
  Other Names: Open surgery
  Groups: Open Rectal Surgery

SUMMARY:
Retrospective cohort study used to analyze trends in minimally invasive versus open surgery in colorectal surgery, over time, in outcome in the laparoscopic, robotic and open surgery groups in patients receiving colorectal resections. Analysis will be performed using data collected through the American College of Surgeons (ACS) National Surgical Quality Improvement Project (NSQIP) database, a national database with deidentified data entered by trained nurse data reviewers.

DETAILED DESCRIPTION:
Perioperative outcomes in patients undergoing laparoscopic compared to open surgery have been improving, and adoption of these procedures has rapidly escalated. Despite this, minimally invasive surgery in rectal cancer is more controversial now than ever before. While laparoscopy was initially limited to non-oncologic operations, it has been shown to produce equivalent oncologic outcomes as open surgery and is now a preferred technique for colon cancer resection. However, laparoscopy is technically challenging in the deep pelvis, and there is concern for adequate resection of rectal cancers.

Multiple clinical trials are ongoing to assess long-term oncologic outcomes in patients with laparoscopically-resected rectal cancers (ACOSOG, ALaCaRT, COLOR II, COREAN)1-4; yet, current data examining perioperative outcomes in these patients is limited.5,6 As there are conflicting conclusions between ongoing randomized control trials about the appropriateness of laparoscopic surgery for rectal cancers, knowledge about perioperative outcomes and trends in these outcomes over time may give surgeons more information to make clinical decisions. To address this gap, the American College of Surgeons (ACS) National Surgical Quality Improvement Program (NSQIP) database was examined to determine the prevalence of laparoscopic surgery and 30-day outcomes over a ten-year period in patients undergoing open and laparoscopic surgery for rectal cancer.

Using the ACS-NSQIP database from 2005-2016, resections for rectal cancer will be studied. The proportion of laparoscopic versus open surgeries performed will be determined by year, and 16 30-day outcomes will be studied in each group. Outcomes include: death, cardiac arrest, cerebrovascular accident, myocardial infarction, pulmonary embolism, venous thromboembolism, pneumonia, prolonged ventilation, superficial or deep incisional surgical site infection, organ space infection, renal insufficiency, acute renal failure, urinary tract infection, length of hospital stay, and operating room time. Multiple logistic regression will be utilized to determine the association between laparoscopic and open technique as well as odds of outcome over time.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Rectal Cancer

Exclusion Criteria:

* Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18+ undergoing surgery for primary diagnosis of rectal cancer between 2005-2016 in the American College of Surgeons National Surgical Quality Improvement Program
Sampling Method: Non-Probability Sample
Enrollment: 31795 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | Post-procedure through day 30
  Outcomes include: death, cardiac arrest, cerebrovascular accident, myocardial infarction, pulmonary embolism, venous thromboembolism, pneumonia, prolonged ventilation, superficial or deep incisional surgical site infection, organ space infection, renal insufficiency, acute renal failure, urinary tract infection, length of hospital stay, and operating room time

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Davis, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No
The ACS-NSQIP database is available by researcher request to the American College of Surgeons. The investigators in this study do not have the authority to share this data independently.

REFERENCES:
- [Background] Fleshman J, Branda M, Sargent DJ, Boller AM, George V, Abbas M, Peters WR Jr, Maun D, Chang G, Herline A, Fichera A, Mutch M, Wexner S, Whiteford M, Marks J, Birnbaum E, Margolin D, Larson D, Marcello P, Posner M, Read T, Monson J, Wren SM, Pisters PW, Nelson H. Effect of Laparoscopic-Assisted Resection vs Open Resection of Stage II or III Rectal Cancer on Pathologic Outcomes: The ACOSOG Z6051 Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1346-55. doi: 10.1001/jama.2015.10529. PMID 26441179
- [Background] Stevenson AR, Solomon MJ, Lumley JW, Hewett P, Clouston AD, Gebski VJ, Davies L, Wilson K, Hague W, Simes J; ALaCaRT Investigators. Effect of Laparoscopic-Assisted Resection vs Open Resection on Pathological Outcomes in Rectal Cancer: The ALaCaRT Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1356-63. doi: 10.1001/jama.2015.12009. PMID 26441180
- [Background] Bonjer HJ, Deijen CL, Haglind E; COLOR II Study Group. A Randomized Trial of Laparoscopic versus Open Surgery for Rectal Cancer. N Engl J Med. 2015 Jul 9;373(2):194. doi: 10.1056/NEJMc1505367. No abstract available. PMID 26154803
- [Background] Jeong SY, Park JW, Nam BH, Kim S, Kang SB, Lim SB, Choi HS, Kim DW, Chang HJ, Kim DY, Jung KH, Kim TY, Kang GH, Chie EK, Kim SY, Sohn DK, Kim DH, Kim JS, Lee HS, Kim JH, Oh JH. Open versus laparoscopic surgery for mid-rectal or low-rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): survival outcomes of an open-label, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jun;15(7):767-74. doi: 10.1016/S1470-2045(14)70205-0. Epub 2014 May 15. PMID 24837215
- [Background] Greenblatt DY, Rajamanickam V, Pugely AJ, Heise CP, Foley EF, Kennedy GD. Short-term outcomes after laparoscopic-assisted proctectomy for rectal cancer: results from the ACS NSQIP. J Am Coll Surg. 2011 May;212(5):844-54. doi: 10.1016/j.jamcollsurg.2011.01.005. Epub 2011 Mar 16. PMID 21414814
- [Background] Jiang JB, Jiang K, Dai Y, Wang RX, Wu WZ, Wang JJ, Xie FB, Li XM. Laparoscopic Versus Open Surgery for Mid-Low Rectal Cancer: a Systematic Review and Meta-Analysis on Short- and Long-Term Outcomes. J Gastrointest Surg. 2015 Aug;19(8):1497-512. doi: 10.1007/s11605-015-2857-5. Epub 2015 Jun 4. PMID 26040854
- [Background] Vargas GM, Sieloff EP, Parmar AD, Tamirisa NP, Mehta HB, Riall TS. Laparoscopy decreases complications for obese patients undergoing elective rectal surgery. Surg Endosc. 2016 May;30(5):1826-32. doi: 10.1007/s00464-015-4463-8. Epub 2015 Aug 19. PMID 26286013
- [Background] Pigazzi A, Ellenhorn JD, Ballantyne GH, Paz IB. Robotic-assisted laparoscopic low anterior resection with total mesorectal excision for rectal cancer. Surg Endosc. 2006 Oct;20(10):1521-5. doi: 10.1007/s00464-005-0855-5. Epub 2006 Aug 1. PMID 16897284